CLINICAL TRIAL: NCT02249104
Title: Epiduo® (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% Pump, Cetaphil® DermaControl™ Moisturizer SPF 30, and Cetaphil® DermaControl™ Foam Wash Regimen in Student Athletes With Mild to Moderate Acne Vulgaris
Brief Title: A Treatment Regimen for Student Athletes With Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10302
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2016-05-26 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2016-04

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene; Adapalene, Benzoyl Peroxide Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acne treatment (Experimental): Adapalene/benzoyl peroxide gel, 0.1%/2.5%, once daily
  Cetaphil Acne Regimen:
  Cetaphil® DermaControl™ Moisturizer SPF 30, once daily and additionally 15 minutes prior to participation in outdoor sports if more than 2 hours elapsed since morning application
  Cetaphil® DermaControl™ Foam Wash, at least twice daily
  Interventions: Drug: Adapalene/benzoyl peroxide gel, 0.1%/2.5%; Other: Cetaphil Acne Regimen

INTERVENTIONS:
Drug: Adapalene/benzoyl peroxide gel, 0.1%/2.5% — Topical AV therapy
  Other Names: Epiduo
Other: Cetaphil Acne Regimen — Cleanse, Moisturize, and Protect
  Other Names: Cetaphil DermaControl Foam Wash; Cetaphil DermaControl Moisturizer SPF 30

SUMMARY:
The goal of this study is to evaluate a complete topical acne regimen consisting of a prescription acne medication (Epiduo® Gel) and an acne-specific cleanser (Cetaphil® DermaControl™ Foam Wash) and moisturizer with sunscreen (Cetaphil® DermaControl™ Moisturizer SPF 30) for safety, efficacy and patient satisfaction in student athletes with acne vulgaris.

DETAILED DESCRIPTION:
The overall purpose of this study was to demonstrate lesion count reduction from baseline, subject satisfaction, and compliance with a regimen of adapalene BPO used in conjunction with a foam wash and moisturizer with sunscreen in student athletes. The study hypothesis was that this regimen would reduce total lesion count (inflammatory and noninflammatory) relative to baseline. The objective of this study was to evaluate the change in lesion count (total, inflammatory, and noninflammatory) in subjects using the CoMMPlete regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females aged 12 years and older who are actively participating in one of 14 Texas University Interscholastic League (UIL) sanctioned athletic activities at the baseline visit (Baseball; Basketball; Cross Country; Football; Golf; Soccer; Softball; Swimming and Diving; Team Tennis; Tennis; Track and Field; Volleyball; and Wrestling).
2. Subjects who agree to be photographed at each visit.
3. Diagnosed with acne vulgaris by a BCD and eligible for treatment with Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5% per PI.
4. Female subjects must have a negative urine pregnancy test (UPT) at Baseline/Visit 1, must be willing to have this test performed at the clinic, and must agree to practice one form of effective methods of non-hormonal contraception for the duration of the study which include: abstinence, IUD (inserted 30 days prior to baseline), double-barrier method, bilateral tubal ligation, or vasectomized partner (at least 90 days prior to baseline).
5. A minimum of 20 but not more than 50 inflammatory (papules and pustules) lesions on the face (excluding the nose) and a minimum of 30 but not more than 100 noninflammatory lesions (open comedones and closed comedones) on the face (excluding the nose).
6. Agree to use the provided study products as their only acne treatment, facial wash and facial moisturizer for the duration of the study.
7. Agree to refrain from temporary and permanent tattoos, paint, or other facial art (including, but not limited to piercings), cosmetic procedures and devices (including, but not limited to facial peels, microdermabrasion and Clarisonic®) on the face for the duration of the study.
8. Subjects aged 12-17 must be willing to read and provide written informed consent/assent in conjunction with a parent/legal guardian who is able and willing to read and provide written consent prior to any study related procedure or subjects aged 18 and older must be willing to read and provide written informed consent prior to any study related procedures.
9. Subjects apprised of the Health Insurance Portability and Accountability Act of 1996 (HIPAA) and applicable state Bill of Rights and are willing to share personal information and data, as verified by signing a written authorization at Screening.
10. Subjects must be willing and able to attend study visits and fulfill dosing requirements.
11. Subjects able to follow study instructions and likely to complete all required visits. In particular, subjects must agree to adhere to the visit schedule and be compliant with the treatment regimen.

Exclusion Criteria:

1. Subjects with nodules and cysts.
2. Female subjects who are pregnant, nursing or planning a pregnancy during the study.
3. Subjects with facial hair, abnormal pigmented vascular skin lesions, abnormal skin pigmentation, or body art (tattoos, permanent or temporary) on the face, which could interfere with subsequent evaluations of dermal responsiveness.
4. Subjects with any systemic or dermatological disorder, a known history of allergies or other medical conditions, which in the opinion of the principal investigator/BCD, could interfere with the conduct of the study, interpretation of results or increase the risk of adverse reactions.
5. Subjects with any known allergies to any of the ingredients listed on the study product labels (refer to study product"s PI and/or current labelling).
6. Subjects who have participated in another interventional, investigational drug or device research study within 30 days of enrollment.
7. Study site staff or sponsor staff, relatives of site staff or sponsor, or other individuals who would have access to the clinical study protocol.
8. Subjects with a washout period less than 1 week for over-the-counter topical acne treatments (with active ingredients such as Benzoyl Peroxide, Salicylic Acid, Sulfur and Resorcinol), prescription topical acne treatment and topical corticosteroids, and use of cosmetic devices (such as Clarisonic® or similar) and less than 4 weeks for topical retinoids.
9. Subjects with a washout period less than 4 weeks for systemic prescription acne treatment and systemic corticosteroids and less than 24 weeks for oral retinoids.
10. Subjects with current sunburn, eczema, atopic dermatitis, perioral dermatitis, rosacea, or other topical conditions on the area to be treated.
11. Subjects who are at risk in terms of precautions, warnings, and contra-indications (refer to the study product"s PI and current labelling).
12. Subjects who foresee unprotected and intense UV exposure during the study (mountain sports, UV radiation, sunbathing, etc.).
13. Subjects with any visible skin condition or facial hair that could interfere with the evaluations.
14. Subjects taking or planning to take topical or systemic medications to treat acne during the course of the study.
15. Subjects taking other medications, supplements, or non-prescription treatments that, in the opinion of the principal investigator/BCD, could interfere with the test results including any regimen of steroidal/non-steroidal anti-inflammatory drugs, or antihistamines, or anabolic steroids.
16. Subjects currently under the treatment for asthma or diabetes (insulin-dependent only).
17. Subjects with planned surgical or cosmetic procedures of the face during the course of the study.
18. Subjects with a history of procedures such as microdermabrasion, chemical peels, intense pulsed light, fillers, Botox®, lasers, photodynamic therapy, red and blue light therapy, etc. in the last 90 days.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-08; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Lain, MD, Principal Investigator — Pflugerville Dermatology Clinical Research
Locations (1):
- Pflugerville Dermatology Clinical Research, Pflugerville, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject, first visit: 20 Aug 2014; Single center study
Groups:
- Acne Treatment: Adapalene/benzoyl peroxide gel, 0.1%/2.5%, once daily
  Cetaphil Acne Regimen:
  Cetaphil® DermaControl™ Moisturizer SPF 30, once daily and additionally 15 minutes prior to participation in outdoor sports if more than 2 hours elapsed since morning application
  Cetaphil® DermaControl™ Foam Wash, at least twice daily
  Adapalene/benzoyl peroxide gel, 0.1%/2.5%: Topical AV therapy
  Cetaphil Acne Regimen: Cleanse, Moisturize, and Protect
Period: Overall Study
Arm/Group | Acne Treatment
Started | 28
Completed | 25
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 27
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Total Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Lesions counted
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Lesions counted | -26.9 (25.3)

2. Secondary Outcome: Percent Change From Baseline in Total Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Percent change | -29.6 (26.9)

3. Secondary Outcome: Mean Change From Baseline in Inflammatory Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Lesions counted
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Lesions counted | -10.8 (9.1)

4. Secondary Outcome: Mean Change From Baseline in Non-inflammatory Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Lesions counted
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Lesions counted | -16.3 (20.5)

5. Secondary Outcome: Percent Change From Baseline in Inflammatory Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Percent change | -35.7 (29.9)

6. Secondary Outcome: Percent Change From Baseline in Non-inflammatory Lesion Count
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acne Treatment
Number analyzed (Participants) | 28
Percent change | -27.1 (34.4)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Acne Treatment
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 18/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acne Treatment (N=28)
Erythema (Skin and subcutaneous tissue disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 5 (5)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Application site pain (General disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
External ear cellulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Immune system disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Open label study with small sample size

Short duration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish, present, or use any results that do not disclose any confidential information furnished by Galderma. The investigator shall provide their draft of such publication to sponsor for review and approval at least 45 days prior to the date of the intended publication. Upon written request from Galderma, within the forty-five (45) day review period, the investigator will delay the publication or presentation for a maximum of an additional one-hundred eighty (180) days.